CLINICAL TRIAL: NCT00954967
Title: Community Intervention Trial for Smoking Cessation With Intensive Advice in Diabetic Patients in Primary Health Care
Brief Title: Trial for Tobacco Cessation With Intensive Advice in Diabetic Patients: the ITADI Project
Acronym: ITADI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Institut Catala de Salut (Other Government); Consorci Sanitari de Terrassa (Other)
Responsible Party: Principal Investigator, USR Metropolitana Nord, Doctor, Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI08/90345
Record Dates: First submitted 2009-08-06; First posted 2009-08-07 (Estimated); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Diabetes Mellitus; Smoking Cessation
Keywords: Diabetes Mellitus; Smoking Cessation; Primary Health Care; Motivational Interview
MeSH Terms: conditions — Diabetes Mellitus; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual care (No Intervention): The subjects in the control group will receive the usual care for smoking cessation in diabetic smokers.
- Lifestyle Counseling (Experimental): The intervention is based on lifestyle advice, motivational interviewing and the use of medications, using the Clinical Practice Guidelines of the Catalan Institute of Health. Health professionals in the intervention group receive a training on the abovementioned techniques.
  Interventions: Behavioral: Lifestyle Counseling

INTERVENTIONS:
Behavioral: Lifestyle Counseling — The intervention is based on lifestyle advice, motivational interviewing and the use of medications, using the Clinical Practice Guidelines of the Catalan Institute of Health. Health professionals in the intervention group receive a training on the abovementioned techniques.
  Arms: Lifestyle Counseling

SUMMARY:
This study addresses an important problem in public health, smoking in diabetics. The morbidity and mortality observed in diabetics is linked to macro and microvascular problems. The consumption of tobacco has a multiplying effect on these vascular problems in diabetics. This study aims to evaluate the effectiveness of an intensive intervention in tobacco addiction in diabetic patients in primary care.

DETAILED DESCRIPTION:
Other objectives of the study are:

1. To study the effectiveness of an intensive smoking cessation intervention in the evolution of the phases of change, as based on the Prochaska and DiClemente model, in diabetic patients attended in primary care.
2. To evaluate the effectiveness of an intensive smoking cessation intervention in the evolution of tabacco consumption in diabetic patients attended in primary care.
3. To quantify the time spent in the intensive smoking cessation intervention compared with the usual care in primary care.

ELIGIBILITY:
Inclusion Criteria:

* diabetic patients who are active smokers
* over the age of 14
* receive routine care in their respective health center

Exclusion Criteria:

* patients with communication difficulties (cognitive deterioration, language barrier)
* patients who normally receive their habitual care in a different health center
* patients with terminal diseases, psychiatric diseases that are unstable, or with addictions to other substances
* patients that are already receiving treatment to quit smoking at the time of recruitment
* patients that are difficult to locate during the study period
* patients that refuse to participate in the study

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 722 (Actual)
Dates: Start 2009-09 (Actual); Primary Completion 2011-01 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Smoking abstinence: Self reported abstinence (6 or more months without smoking) confirmed by an expired air carbon monoxide concentration of 6 parts per millions or less | 12 months after initiation of study

SECONDARY OUTCOMES:
Evolution of the phases of change of the Prochaska and DiClemente model | 12 months after initiation of the study
Number of cigarettes per day | 12 months after initiation of the study
Total time (minutes) spent in the intensive smoking cessation intervention | 12 months after initiation of the study

CONTACTS AND LOCATIONS:
Overall Officials: Santiago Pérez, MD, Principal Investigator — CAP La Llagosta
Locations (1):
- IDIAP Jordi Gol, Barcelona, Spain

REFERENCES:
- [Derived] Roig L, Perez S, Prieto G, Martin C, Advani M, Armengol A, Roura P, Manresa JM, Briones E; ITADI Study Group. Cluster randomized trial in smoking cessation with intensive advice in diabetic patients in primary care. ITADI Study. BMC Public Health. 2010 Feb 4;10:58. doi: 10.1186/1471-2458-10-58. PMID 20132540